CLINICAL TRIAL: NCT05278156
Title: Phase II, Double Blind, Randomized, Placebo Controlled, Parallel Group, Trial to Explore Efficacy, Safety and Pharmacokinetics of CPL500036 (PDE10A Inhibitor) in Patients With an Acute Exacerbation of Schizophrenia
Brief Title: Efficacy, Safety and Pharmacokinetics Study of CPL500036 (PDE10A Inhibitor) in Patients With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celon Pharma SA (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02PDE2019
Record Dates: First submitted 2022-02-09; First posted 2022-03-14 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPL500036 low dose (Experimental): Patients are to receive 20 mg of CPL500036 administered once dail for 28-days treatment period.
  Interventions: Drug: CPL500036 - low dose
- CPL500036 high dose (Experimental): Patients are to receive 40 mg of CPL500036 administered once dail for 28-days treatment period.
  Interventions: Drug: CPL500036 - high dose
- Placebo (Placebo Comparator): Patients are to receive placebo administered once dail for 28-days treatment period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CPL500036 - low dose — CPL500036 is to be oral administered. Each patient is to take 2 capsules with active substance and 2 capsules of placebo daily.
  Arms: CPL500036 low dose
Drug: CPL500036 - high dose — CPL500036 is to be oral administered. Each patient is to take 4 capsules with active substance daily.
  Arms: CPL500036 high dose
Drug: Placebo — Placebo is to be oral administered. Each patient is to take 4 capsules of placebo daily.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy, safety, tolerability and pharmacokinetics (PK) properties of CPL500036 compound (PDE10a inhibitor) in patients with an acute exacerbation of schizophrenia after 28 days of administration..

DETAILED DESCRIPTION:
This is a double-blind, randomized, placebo controlled, parallel group, dose ranging study to explore the efficacy, safety, tolerability and PK of 2 different doses of CPL500036 (phosphodiesterase 10A [PDE10A] inhibitor) in patients with an acute exacerbation of schizophrenia. Approximately 165 patients will be randomized at a 1:1:1 ratio and will be dosed with 20 mg CPL500036, 40 mg CPL500036 or placebo once daily for 28 consecutive days (Day 1 to Day 28). Patients will remain in house for the duration of the Treatment Period. The study will comprise of a Screening Period (that will include a prior Medication Washout Period), a Treatment Period and a Follow-up Period. After discharge from the Clinical Unit, patients will return to the Clinical Unit for 2 once weekly Follow-up Visits. Approximately 30% of the patients (17 patients in each of the 3 treatment groups) will undergo extensive PK sampling during the Treatment Period, and the remaining 70% of the patients will only undergo sparse PK sampling.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a primary diagnosis of schizophrenia confirmed by clinical interview [SCID-5-CT].
2. Male or female patient aged 18 to 65, inclusive, at Screening.
3. The patient's with exacerbation of psychotic symptoms
4. The patient has a score of 5 or higher in 3 or more items of the following PANSS items at Screening and Baseline
5. The patient has a PANSS Total Score of 80 or higher during Screening and on Baseline
6. The patient of childbearing potential willing to use acceptable forms of contraception.
7. The patient has a score in CGI-S scale of 4 or greater at Screening and on Baseline
8. The patient is able to and agrees to remain off prior antipsychotic medication and all excluded medications as outlined in the protocol for the duration of the Treatment Period.
9. The patient is able to sign informed consent after receiving information about the trial and has the ability and willingness to comply with the requirements and restrictions of the study protocol.

Exclusion Criteria:

1. The patient has a decrease in the PANSS Total Score at Baseline compared with the Total Score at Screening.
2. Patient who recently participated in another interventional clinical study with an Investigational Medicinal Product.
3. The patient has uncontrolled abnormality which may impact the ability of the patient to participate or potentially confound the study results.
4. The patient has a history of severe head injury, traumatic brain injury, myocardial infarction or stroke.
5. The patient has a moderate or severe substance use disorder for alcohol or other substances of abuse except nicotine or caffeine.
6. The patient is pregnant or lactating or intending to become pregnant or intending to donate ova.
7. The patient has a history of or known personality disorder or other psychiatric disorder that, in the opinion of the Investigator, would interfere with participation in the study.
8. The patient is considered by the Investigator to be at imminent risk of suicide or injury to self or others.
9. The patient has chronic movement disorder that may interfere with the interpretation of study results.
10. The patient has any existing or previous history of cancer or has newly diagnosed diabetes.
11. The patient has long QT syndrome or is under treatment with antiarrhythmic drugs.
12. The patient is considered to be treatment resistant. .
13. The patient has received electroconvulsive therapy.
14. The patient has any laboratory values outside the normal range that are considered by the Investigator to be clinically significant at Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline in PANSS positive subscale at Day 28. | Day -1, Day 28
  The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient.Total score is 210 points. The higher PANSS total score, the more severe schizophrenia.

SECONDARY OUTCOMES:
Change from baseline in PANSS positive subscale at Week 1, 2 and 3 | Day -1, Week 1, 2 and 3
  The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient.Total score is 210 points. The higher PANSS total score, the more severe schizophrenia.
Change from baseline in PANSS Total Score at Weeks 1, 2, 3, 4 | Day -1, Week 1, 2, 3 and 4
  The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient.Total score is 210 points. The higher PANSS total score, the more severe schizophrenia.
Change from Baseline in PANSS Subscales Using the Marder 5 factor Model at Weeks 1, 2, 3, and 4 | Day -1, Week 1, 2, 3 and 4
  The PANSS is a 30-item scale used to measure symptoms of schizophrenia.
Change from Baseline in PANSS Negative Subscales at Weeks 1, 2, 3 and 4 | Day -1, Week 1, 2, 3 and 4
  The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient.Total score is 210 points. The higher PANSS total score, the more severe schizophrenia.
Change from Baseline in PANSS general psychopathology Subscale at Weeks 1, 2, 3 and 4 | Day -1, Week 1, 2, 3 and 4
  The PANSS is a 30-item scale used to measure symptoms of schizophrenia. The scale has 7 positive symptom items, 7 negative symptom items, and 16 general psychopathology symptom items. Each item is scored on a 7-point scale by the clinical rater based on a clinical interview with the patient.Total score is 210 points. The higher PANSS total score, the more severe schizophrenia.
Percentage of Clinical Responders Based on the PANSS Total Score. | Day -1, Week 1, 2, 3 and 4
  Clinical responder is defined as a ≥ 30% decrease from baseline.
Change from Baseline in Clinical Global Impression Severity (CGI-S) Score at Weeks 1, 2, 3, and 4 | Day -1, Week 1, 2, 3 and 4
  CGI-S scale is a physician-rated scale that is designed to rate the severity of the patient's illness at the time of assessment. It is a 7-point assessment where 1= normal (not at all ill) and 7 = among the most extremely ill patients.
Clinical Global Impression Scale Improvement (CGI-I) Score at Weeks 1, 2, 3, 4. | Day -1, Week 1, 2, 3 and 4
  CGI-I is a 7 points scale that requires the clinician to assess how much the patient's illness has improved or worsened during treatment. It is a 7-point assessment where 1= Very much improved and 7 = Very much worse
Change from Baseline in Brief Assessment of Cognition in Schizophrenia (BACS) Score at Weeks 2 and 4. | Day -1, Week 2 and 4
  BACS is specifically designed to measure treatment-related improvements in cognition. The BACS is a cognition assessment battery that assesses 6 domains of cognitive function found to be consistently impaired in schizophrenia: verbal memory, working memory, motor speed, attention, executive functions, and verbal fluency.
Number of abnormal clinically significant values in vital signs (heart rate, blood pressure, respiratory rate) results. | up to 6 weeks
Number of abnormal clinically significant findings in electrocardiogram results. | up to 6 weeks
  The following electrocardiogram parameters will be assess: PR interval, QRS interval, RR interval, QT interval and QTc interval.
Number of abnormal clinically significant values in laboratory tests (hematologic, clinical chemistry, coagulation and urinalysis) results. | up to 6 weeks
Number of abnormal physical, neurological, ophthalmological and dermatological examination findings. | up to 6 weeks
Number and intensity of extrapyramidal side effects. | up to 6 weeks
  It will be assessed by using Extrapyramidal Symptom Rating Scale (ESRS). This scale is using to assess four types of drug-induced movement disorders (DIMD): Parkinsonism, akathisia, dystonia, and tardive dyskinesia.
Number of adverse events. | up to 6 weeks
  All adverse events that occurence during study will be assessed.
CPL500036 Cmax - Maximum observed concentration | up to 24 hours after administration on Day 7
CPL500036 Tmax - Time corresponding to occurrence of Cmax | up to 24 hours after administration on Day 7
CPL500036 AUC (0-24h) - Area under the curve from time zero to 24 hours | up to 24 hours after administration on Day 7
CPL500036 AUC T1/2 - Apparent terminal elimination half-life | up to 24 hours after administration on Day 7
CPL500036 CL/F (Apparent clearance) and Vz/F (apparent volume of distribution during terminal phase) | up to 24 hours after administration on Day 7
CPL500036 Cthrough - Concentration immediately prior to dosing | up to 24 hours after administration on Day 7

CONTACTS AND LOCATIONS:
Locations (16):
- Hungary (5):
  - Department of Psychiatry and Psychotheraapy of Semmelweis University, Budapest
  - Semmelweis University, Faculty of Medicine, Department of Psychiatry and Psychotherapy, Budapest
  - Department of Psychiatry, Mental hygiene and Addictology of Petz Aladár County Teaching Hospital, Győr
  - Bács-Kiskun County Teaching Hospital Kalocsa Holy Cross Hospital, Kalocsa
  - Psychiatry Department of Tolna County Balassa Janos Hospital, Szekszárd
- Poland (4):
  - Uniwersytecki Szpital Kliniczny, Bialystok
  - Wojewódzki Szpital dla Nerwowo i Psychicznie Chorych, Bolesławiec
  - Samodzielny Publiczny Psychiatryczny Zakład Opieki Zdrowotnej, Choroszcz
  - Wojewódzki Szpital dla Psychicznie i Nerwowo Chorych, Gmina Świecie
- Ukraine (7):
  - Ivano-Frankivsk National Medical University, Department of Psychiatry, Narcology and Medical Psychology, Ivano-Frankivsk
  - Communal non-profit enterprise "Clinical Hospital "PSYCHIATRY"" of the executive body of the Kyiv City Council (Kyiv City State Administration), Center for Primary Psychotic Episode and Modern Treatment Methods., Kyiv
  - Communal non-commercial enterprise of the Kyiv Regional Council "Regional Psychiatric-Narcological Medical Association", women's department No. 2, men's department No. 10., Kyiv
  - Communal non-commercial enterprise of the Lviv Regional Council "Lviv Regional Clinical Psychoneurological Dispensary",, Lviv
  - Communal non- commercial enterprise of Lviv Regional Council "Lviv Regional Clinical Psychiatric Hospital",, Lviv
  - Ternopil National Medical University named after I.Y. Gorbachevskiy of the Ministry of Health of Ukraine, Department of Psychiatry, Narcology and Medical Psychology, Ternopil
  - Vinnytsia National Medical University named after M.I. Pirogov, Department of Psychiatry, Narcology and Psychotherapy with a course of postgraduate education, Vinnytsia

DOCUMENTS (2):
  • Study Protocol (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT05278156/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/56/NCT05278156/SAP_001.pdf